CLINICAL TRIAL: NCT02775981
Title: A Phase-1 Study Comparing the Pharmacokinetics of Intranasal RX0041-002 in Hepatic-Impaired Individuals and Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetic Study of Intranasal RX0041-002 in Hepatic-Impaired Individuals and Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Project Solutions, Inc. (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTS2015014
Record Dates: First submitted 2016-03-23; First posted 2016-05-18 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Analgesic Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): RX0041-002
  Interventions: Drug: RX0041-002

INTERVENTIONS:
Drug: RX0041-002

SUMMARY:
The primary objective of this study is to evaluate the potential effect of hepatic impairment on the systemic pharmacokinetics of RX0041-002 following single dose intranasal administration. The secondary objective is to evaluate the safety and tolerability of intranasal RX0041-002 in subjects with normal hepatic function and hepatic impairment.

DETAILED DESCRIPTION:
This is a Phase 1, single dose, open-label study comparing the plasma pharmacokinetics and safety of RX0041-002 between subjects with hepatic impairment and age/gender/BMI-matched subjects with normal hepatic function.

DOSAGE

All subjects will receive a single treatment consisting of four (4) ml of a 4% solution of RX0041-002 (corresponding to 160 mg cocaine HCl) applied for 20 minutes to both nostrils using cotton pledgets. RX0041-002 Topical Solution (4%) will be provided by the Sponsor, supplied in 4 mL bottles. RX0041-002 Topical Solution contains citric acid, D&C Yellow No. 10, FD&C Green No. 3, sodium benzoate, and water.

DURATION OF STUDY

Total duration of study participation for each subject will be approximately 23 days not counting the variable 30 days for adverse event follow-up and resolution, if required. During that time, subjects will be screened for a maximum of 21 days and then confined to the study unit for approximately 45 hours for Day -1 evaluations, dosing (Day 1), blood sampling and safety assessments (Day 1-2).

NUMBER OF SUBJECTS

A sufficient number of subjects will be enrolled to complete 12 subjects with hepatic impairment, male or female volunteers ≥ 18 years of age. An additional 12 healthy, non-hepatically impaired, male or female volunteers will be enrolled as the comparator group. These subjects will be approximately age, body mass index (BMI) & gender-matched to the subjects with hepatic impairment. Hepatic impairment will be classified as moderate or severe and each grade/class will be defined according to Child-Pugh classification (Class B or C) . The liver impairment will be identified by a typical medical history, physical examination, coagulation and abnormal liver function tests (including bilirubin and albumin) at screening.

SAFETY PARAMETERS

Prior to enrollment (screening) and at the completion of the study, or at premature discontinuation, each subject will undergo a complete physical examination plus vital signs, clinical laboratory testing (serum chemistry, hematology, and urinalysis), and coagulation. In addition, subjects will be screened for inclusion with a 12-lead electrocardiogram, a urinary screen for drugs of abuse and blood tests for alcohol, serology tests for HIV antibody. Breath alcohol and urine drug screens will be repeated at check-in on Day -1 of the study. Females of child bearing potential will also be screened for inclusion with a serum pregnancy test. Urine pregnancy tests will also be performed at check-in on Day -1.

Each subject will be queried for the occurrence of adverse experiences following dosing and during blood sampling. Vital sign monitoring and recordings, will be obtained at baseline (pre-dose) (Day 1). Blood pressure, heart rate, respiratory rate and oral temperature will be taken and recorded every 15 minutes beginning immediately prior to dosing and for every 15 minutes for the first 60 minutes following pledget insertion. For the next 120 minutes (up to 180 minutes' post pledget insertion) vital sign recordings to include blood pressure, heart rate, respiratory rate and oral temperature measurements will be taken and recorded every 30 minutes to the 180 minute (3 Hour) post pledget insertion time point. Vital sign recordings to include blood pressure, heart rate, respiratory rate and oral temperature measurements will continue to be taken and recorded at hour 4, 6, 8, 10, 12, 16, 20, 24, 28 and 32 hours from time of pledget insertion or if necessary until the patient is clinically stable.

A nasal exam will be conducted, visually, pre-dose (Day 1) and at the end of study (Day 2) to determine if irritation is present at the application site following drug administration.

PHARMACOKINETIC BLOOD SAMPLING AND ANALYSIS

Pharmacokinetic blood samples will be drawn at the following times relative to the initiation of RX0041-002 dosing.

Subjects will be dosed and blood pharmacokinetic sampling will be conducted at 0 hour (pre-dose), and post dose at: 7 minutes, 15 minutes, 20 minutes, (immediately after pledget removal) 30 minutes, 45 minutes, 60 minutes, 75 minutes, 90 minutes, 105 minutes, and 2, 3, 4, 6, 8, 10, 12, 24, 28 and 32 hours, based upon the beginning of dose application. For each time point, a minimum of 8 ml of blood will be sampled.

Total concentrations of cocaine and it major metabolites will be determined in all samples.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Greater than or equal to 18 years of age and able to understand and comply with protocol requirements, provide written informed consent and HIPAA authorization; ± 10 years for individual age-matched controls.
3. Females (if of child-bearing potential and sexually active) and males (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method from the first dose and for 8 days following administration of study drug. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm, intrauterine device (IUD), condom, surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method or withdrawal.
4. BMI ≥ 18 ≤ 32 ; ± 20% for BMI-matched controls
5. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance.
6. In general, good health aside from hepatic disease (for the hepatically impaired group only) and associated conditions as ascertained by physical examination (PE) including measurement of supine and standing vital signs, medical history, clinical laboratory evaluation, and 12-lead electrocardiogram (ECG).

   Hepatic Subjects
7. Hepatic-impaired subjects will be Class B or C according to Child-Pugh classification. The hepatic impairment will have been identified by a typical medical history, physical examination, coagulation tests and abnormal liver function tests (including bilirubin and albumin) at screening.

   Healthy Volunteers
8. Volunteers will be healthy and age, BMI and gender-matched controls for the hepatic subjects.

Exclusion Criteria:

A subject will be excluded from the study if he or she meets the following criteria:

1. Less than 18 years of age.
2. Has a known allergy to any ester based anesthetics including cocaine HCl, procaine, tetracaine, chloroprocaine, dibucaine, or benzocaine amide based anesthetic allergies are NOT exclusionary. Amide based anesthetics are : lidocaine, mepivicaine, bupivicaine, levobupivicaine, ropivicaine, etidocaine, prilocaine, and articaine.
3. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study.
4. The use of amphetamines, methylphenidate or other stimulant prescription and nonprescription products such as pseudoephedrine, bronchial inhalers containing sympathomimetics (epinephrine or other beta-receptor agonist) or herbal products in the 7 days prior to screening or has a need to use these drugs during the course of the study.
5. Use of any Seratonin uptake inhibitor/Serotonin-norepinephrine reuptake inhibitors, antidepressants or tricyclic antidepressant up to7 days or 5 half-lives (whichever is longer) prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
6. Use of Monoamine Oxidase Inhibitor drugs up to 14 days prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
7. GI abnormalities
8. History of hepatitis (for healthy control subjects only)
9. Elevated aspartate aminotransferase/alanine aminotransferase /bilirubin (for healthy control subjects only),
10. HIV
11. Excessive use of alcohol/tobacco/caffeine.
12. Has previously received study drug.
13. Has a history of abuse of controlled substances, nasal or otherwise, or has damage to the nasal space, that in the opinion of the investigator might interfere with the ability to absorb RX0041-002.
14. Has severely traumatized mucosa or sepsis in the nasal cavity.
15. Has participated in an investigational study or received an investigational drug within 30 days preceding the randomization.
16. Is a pregnant or nursing mother.
17. Has a positive pregnancy test at Screening or Day -1.
18. Has a history of seizure, with the exception of febrile seizures.
19. Has symptomatic cardiovascular disease.
20. Has a history of or currently suffers from hyperthyroidism.
21. Has a known personal or family history of hereditary pseudocholinesterase deficiency. Study participants will be screened by asking about personal or family history of anesthetic reaction, anesthetic death, and previous diagnosis of psuedocholinesterase deficiency in a relative or personally. Subjects identified with pseudocholinesterase deficiency are at risk for delayed recovery with certain anesthetics (e.g. succinylcholine and ester-based anesthetics).
22. Has a known personal or family history of pheochromocytoma. Study participants will be specifically asked if they have been treated for a pheochromocytoma previously or if they have a family member who has been diagnosed with pheochromocytoma (since 10% of these are familial).
23. Has a known personal or family history of adrenal tumor.
24. Clinically significant ECG abnormalities, based upon the impression of the investigator.
25. Has a positive urine test result for drugs of abuse (amphetamines, barbiturates, cocaine metabolites, opiates and oxycodone) or cannabinoids at Screening or on Day 1; exception for hepatic subjects who may medically require one of the drugs for treatment (e.g., periodic opiates) and may, at the discretion of the investigator, be positive at screening, but must be negative at Day -1.
26. Blood chemistry values judged clinically significant by the investigator. aa.Donation of blood (one pint or greater) within four weeks prior to administration of study medication.

bb. Not suitable for entry into the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cax) | 32 Hours
Area under the plasma concentration versus time curve (AUC) | 32 Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Clinical Researc, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided